CLINICAL TRIAL: NCT01383135
Title: Biodistribution and Safety of the PET Probes [18F]FPRGD2 and [18F]FPPRGD2
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-16118; SU-09022010-6791 (Other: Stanford University); VAR0047 (Other: OnCore Number)
Record Dates: First submitted 2011-05-31; First posted 2011-06-28 (Estimated); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer; Non-Small-Cell Lung Cancer; Glioblastoma; Other Cancers
Keywords: Healthy volunteers
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Healty Volunteers (Other): Normal volunteers to receive 5 to 14 mCi F18-FPPRGD2 by intravenous (IV) injection.
  Interventions: Drug: F18-FPPRGD2
- Breast Cancer (Experimental): Breast cancer patients to receive 4 to 11 mCi F18-FPPRGD2 by IV injection.
  Interventions: Drug: F18-FPPRGD2
- Glioblastoma Multiform (brain) (Experimental): Glioblastoma multiform patients to receive 5 to14 mCi F18-FPPRGD2 by IV injection.
  Interventions: Drug: F18-FPPRGD2
- Lung Cancer (Experimental): Lung cancer patients to receive X to XX mCi F18-FPPRGD2 by IV injection.
  Interventions: Drug: F18-FPPRGD2

INTERVENTIONS:
Drug: F18-FPPRGD2 — Radiopharmaceutical administered for imaging, up to 14 mCi intravenous (IV).

SUMMARY:
The purpose of the study was to conduct a pilot test of new tracers ([18F]FPRGD2 and [18F]FPPRGD2) to define normal tracer biodistribution (where the tracer goes), stability (how much metabolises), pharmacokinetics (how much stays in which organs and for how long), and radiation dosimetry (organ radiation dose). Healthy volunteers provided the normal biodistribution data.

The same radiopharmaceutical was also tested in breast cancer, glioblastoma multiform (brain cancer), and lung cancer.

DETAILED DESCRIPTION:
The tracer [18F]FPRGD2 was not evaluated in this study. The protocol title was never amended to reflect this.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

1. Must be 18 years of age or older.
2. Must have no known medical problems and have had a full medical exam within 6 months of the study.
3. Must understand and voluntarily have signed an Informed Consent after its contents have been fully explained.
4. Women of child bearing potential (as defined as women who are not post menopausal for 12 months or who have had no previous surgical sterilization).
5. Men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation and for 30 days after the last dose.

Cancer subjects:

1. Greater than 18 years-old at the time of radiotracer administration
2. Provides written informed consent
3. Diagnosed with advanced non-small cell lung cancer (NSCLC), breast cancer, pancreatic cancer and glioblastoma multiforme (GBM); patients will undergo bevacizumab or Cyberknife therapy
4. Able to remain still for duration of each imaging procedure (about one hour)

Exclusion Criteria

1. Less than 18 years-old at the time of radiotracer administration
2. Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-10; Primary Completion 2012-04 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Gambhir, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Volunteers: 5 to 14 mCi F18-FPPRGD2 by intravenous (IV) injection.
- Breast Cancer: 4 to 11 mCi F18-FPPRGD2 by IV injection
- Glioblastoma Multiform Patients: 5 to14 mCi F18-FPPRGD2 by IV injection
- Lung Cancer: X to XX mCi F18-FPPRGD2 by IV injection
Period: Overall Study
Arm/Group | Healthy Volunteers | Breast Cancer | Glioblastoma Multiform Patients | Lung Cancer
Started | 6 | 8 | 9 | 4
Completed | 5 | 8 | 8 | 4
Not Completed | 1 | 0 | 1 | 0
Not completed — Not Scanned / Imaged | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Breast Cancer Patients: 4 to 11 mCi F18-FPPRGD2 by IV injection
- Glioblastoma Multiforme: 5 to14 mCi F18-FPPRGD2 by IV injection
- Total: Total of all reporting groups
Arm/Group | Healthy Volunteers | Breast Cancer Patients | Glioblastoma Multiforme | Lung Cancer | Total
Number analyzed (Participants) | 6 | 8 | 9 | 4 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 7 | 3 | 22
  >=65 years | 0 | 2 | 2 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 4 | 2 | 18
  Male | 2 | 0 | 5 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 7 | 8 | 2 | 19
  Unknown or Not Reported | 4 | 1 | 1 | 2 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 5 | 6 | 3 | 2 | 16
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Tracer Dosimetry by Organ
Description: Normal radiopharmaceutical biodistribution was analyzed visually to obtain dosimetry data in healthy volunteers. Organs with the highest radiation absorbed dose (dosimetry) are provided below. Dosimetry was calculated by drawing regions-of-interest around organs with visually appreciable radiopharmaceutical uptake greater than background and using organ-level internal dose assessment software from Vanderbuilt University (2003).
  Results are reported in mSv/MBq (milli-Sieverts per mega-Bequerel) which is a measurement of the mean absorbed radiation dose within an organ.
Time Frame: 5 hours
Population: Per protocol, data were collected for this outcome from the Healthy Volunteers group only, and only those that completed all scans are included.
Measure: Mean (Standard Deviation); unit: mSv/MBq
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 4
mSv/MBq
  Kidneys | 0.3603 (0.1852)
  Liver | 0.0988 (0.0379)
  Bladder | 0.8615 (0.4362)
  Bowel | 0.5290 (0.2364)

2. Primary Outcome: F18-FPPRGD2 Time-activity at Specified Timepoints
Description: Radiopharmaceutical pharmacokinetics describe the change in radiopharmaceutical distribution in the body (from the blood to organs, tissues, cells) over time. Radiopharmaceutical pharmacokinetics are used to determine optimal imaging time, ie, when target activity (organ or cell of interest) is greater than background activity (blood). Optimal imaging time must also be balanced with tracer bio-metabolism and radioactive decay. F18-FPPRGD2 pharmacokinetics was measured in healthy volunteers to estimate optimal imaging time. Scans were used to visually identify regions of interest (organs of F18-FPPRGD2 accumulation), and detected radiation was plotted as a measurement over time.
Time Frame: 30, 60, and 90 minutes post-injection
Population: Per protocol, data were collected for this outcome from the Healthy Volunteers group only. 4/5 volunteers were able to complete all of the scans. 1/5 participant could only complete one of the four scans and was not included in pharmacokinetic calculations.
Measure: Mean (Standard Deviation); unit: Percentage of tracer remaining in blood
Groups:
- Healthy Volunteers: 5-14 mCi IV F18- FPPRGD2: radiopharmaceutical administered for imaging followed by PET/CT scan
Arm/Group | Healthy Volunteers
Number analyzed (Participants) | 4
Percentage of tracer remaining in blood
  30 minutes post-injection | 26 (17)
  60 minutes post-injection | 18 (14)
  90 minutes post-injection | 8 (2)

3. Primary Outcome: Sensitivity of F18-FPPRGD2 PET/CT in Breast Cancer
Description: Sensitivity is the ability of a test to correctly identify patients with the disease being investigated. In this instance, how well F18-FPPRGD2 PET/CT detects true-positive patients. Sensitivity is defined as [TP/ (TP+FN)], where TP= true positive, and FN = false negative. The outcome is reported as a percentage without dispersion. A higher percentage indicates a greater probability that a lesion identified based on scan results is cancerous, and a lower percentage indicates reduced confidence in that result.
Time Frame: 3 hours
Population: Per protocol, data were collected for this outcome from the Breast Cancer Patients group only. In a per-lesion analysis, a total of 30 lesions were evaluated at PET/CT scanning with F18-FPPRGD2.
Measure: Number; unit: percentage of sensitivity
Units Other Than Participants: Lesions
Groups:
- Breast Cancer Patients: 4-11 mCi IV F18- FPPRGD2: radiopharmaceutical administered for imaging followed by PET/CT scan
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 8
Number analyzed (Lesions) | 30
percentage of sensitivity | 95.7

4. Primary Outcome: Specificity of F18 FPPRGD2 PET/CT in Breast Cancer
Description: Specificity is the ability of a test to correctly identify patients who do not have the disease being investigated. In this instance, how well F18 FPPRGD2 PET/CT detects true-negative patients. Specificity is:
  [TN/ (TN+FP)], where TN= true negative, and FP = false positive.
Time Frame: an estimated average of 3 hours
Population: Per protocol, data were collected for this outcome from the Breast Cancer Patients group only. Other cohorts are not included, and the outcome was only assessed in the breast cancer cohort.
Measure: Number; unit: percentage of specificity
Arm/Group | Breast Cancer Patients
Number analyzed (Participants) | 8
percentage of specificity | 100

5. Primary Outcome: Glioblastoma Primary Tumor Response Assessed by PET Scan
Description: Primary tumor response was assessed after 6 weeks of treatment as the change in tumor metabolism based on the maximum standardized uptake value (SUVmax) as determined by positron emission tomography (PET) scans. Decreased SUVmax correlates to a reduction of tumor metabolism, and is considered an indicator of primary tumor response. Reduction of SUVmax was determined as the change from baseline in uptake of F-18FPPRGD2. The outcome is reported as the baseline and week 6 values, with standard deviation.
Time Frame: Baseline and Week 6
Population: Per protocol, data were collected for this outcome from the Glioblastoma Multiforme group only. Participants in the Glioblastoma Multiforme group who completed the imaging schedule were included in the analysis.
Measure: Mean (Standard Deviation); unit: SUVmax
Groups:
- Glioblastoma Multiforme: F18- FPPRGD2: radiopharmaceutical administered for imaging, up to 14 mCi i.v.
Arm/Group | Glioblastoma Multiforme
Number analyzed (Participants) | 6
SUVmax
  Pretreatment | 1.7 (0.6)
  Week 6 | 1.3 (0.5)
Statistical Analysis 1: Comparison: Glioblastoma Multiforme; Comparison made between baseline tumor values and tumor values 6-weeks post-bevacizumab therapy; Test type: Superiority or Other; p = .034, t-test, 2 sided — GraphPad (GraphPad Software, San Diego, Calif) was used for the paired two-sample t test and was performed to compare SUVmax values. P < .05 was considered to indicate a significant difference

6. Secondary Outcome: Glioblastoma Primary Tumor Response Assessed by CT Scan
Description: Primary tumor response was assessed after 6 weeks of treatment as the change in tumor metabolism based on the maximum standardized uptake value (SUVmax) as determined by computed tomography (CT) scans. Decreased SUVmax correlates to a reduction of tumor metabolism, and is considered an indicator of primary tumor response. Reduction of SUVmax was determined as the change from baseline in uptake of F-18FPPRGD2. The outcome is reported as the mean difference from baseline to week 6, with standard deviation.
Time Frame: Baseline and Week 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Glioblastoma Multiforme: F18-FPPRGD2: radiopharmaceutical administered for imaging, up to 14 mCi IV
Arm/Group | Glioblastoma Multiforme
Number analyzed (Participants) | 6
percentage change | -11.0 (80.7)

ADVERSE EVENTS:
Groups:
- Lung Cancer: 5 to14 mCi F18-FPPRGD2 by IV injection
Arm/Group | Healthy Volunteers | Breast Cancer Patients | Glioblastoma Multiforme | Lung Cancer
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/8 | 0/9 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/8 | 0/9 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/8 | 0/9 | 0/4

LIMITATIONS AND CAVEATS:
This study is a pilot study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No